CLINICAL TRIAL: NCT02500953
Title: A Placebo-controlled, Double-blind, Single and Multiple Oral Dose Study and a Treatment Schedule-finding Study in Non-elderly, Healthy Japanese Male and Female Subjects and Caucasian Male Subjects
Brief Title: A Single and Multiple Oral Dose Study and a Treatment Schedule-finding Study in Non-elderly, Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Astellas Pharma Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Triple
Other Study IDs: 3325-CL-0001
Record Dates: First submitted 2015-07-15; First posted 2015-07-17 (Estimated); Last update posted 2015-07-17 (Estimated); Status verified 2015-07

CONDITIONS: Pharmacokinetics of ASP3325 in Non-elderly, Healthy Adult Japanese Male and Female, and Caucasian Male Subjects
Keywords: ASP3325; pharmacokinetics; pharmacodynamics
MeSH Terms: interventions — ASP3325

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (27):
- Japanese male single fasted ASP dose-1 (Experimental): ASP3325 will be administered as a single oral dose with 240 mL of water to subjects who have been fasting from 22:00 on the day before administration.
  Interventions: Drug: ASP3325
- Japanese male single fasted ASP dose-2 (Experimental): ASP3325 will be administered as a single oral dose with 240 mL of water to subjects who have been fasting from 22:00 on the day before administration.
  Interventions: Drug: ASP3325
- Japanese male single fasted ASP dose-3 (Experimental): ASP3325 will be administered as a single oral dose with 240 mL of water to subjects who have been fasting from 22:00 on the day before administration.
  Interventions: Drug: ASP3325
- Japanese male single fasted ASP dose-4 (Experimental): ASP3325 will be administered as a single oral dose with 240 mL of water to subjects who have been fasting from 22:00 on the day before administration.
  Interventions: Drug: ASP3325
- Japanese male single fasted ASP dose-5 (Experimental): ASP3325 will be administered as a single oral dose with 240 mL of water to subjects who have been fasting from 22:00 on the day before administration.
  Interventions: Drug: ASP3325
- Japanese male single fasted ASP dose-6 (Experimental): ASP3325 will be administered as a single oral dose with 240 mL of water to subjects who have been fasting from 22:00 on the day before administration.
  Interventions: Drug: ASP3325
- Japanese male single fasted ASP dose-7 (Experimental): ASP3325 will be administered as a single oral dose with 240 mL of water to subjects who have been fasting from 22:00 on the day before administration.
  Interventions: Drug: ASP3325
- Japanese female single fasted ASP dose-3 (Experimental): ASP3325 will be administered as a single oral dose with 240 mL of water to subjects who have been fasting from 22:00 on the day before administration.
  Interventions: Drug: ASP3325
- Japanese female single fasted ASP dose-5 (Experimental): ASP3325 will be administered as a single oral dose with 240 mL of water to subjects who have been fasting from 22:00 on the day before administration.
  Interventions: Drug: ASP3325
- Caucasian male single fasted ASP dose-3 (Experimental): ASP3325 will be administered as a single oral dose with 240 mL of water to subjects who have been fasting from 22:00 on the day before administration.
  Interventions: Drug: ASP3325
- Caucasian male single fasted ASP dose-5 (Experimental): ASP3325 will be administered as a single oral dose with 240 mL of water to subjects who have been fasting from 22:00 on the day before administration.
  Interventions: Drug: ASP3325
- Japanese male single fed ASP dose-5 (Experimental): ASP3325 will be administered as a single oral dose with 240 mL of water to subjects after a meal.
  Interventions: Drug: ASP3325
- Japanese male single fasted placebo (Experimental): Placebo will be administered as a single oral dose with 240 mL of water to subjects who have been fasting from 22:00 on the day before administration.
  Interventions: Drug: Placebo
- Japanese female single fasted placebo (Experimental): Placebo will be administered as a single oral dose with 240 mL of water to subjects who have been fasting from 22:00 on the day before administration.
  Interventions: Drug: Placebo
- Caucasian male single fasted placebo (Experimental): Placebo will be administered as a single oral dose with 240 mL of water to subjects who have been fasting from 22:00 on the day before administration.
  Interventions: Drug: Placebo
- Japanese male single fed placebo (Experimental): Placebo will be administered as a single oral dose with 240 mL of water to subjects after a meal.
  Interventions: Drug: Placebo
- Japanese male multiple ASP dose-3 (Experimental): ASP3325 will be administered as multiple oral doses with 240 mL of water, three times a day, just after a meal.
  Interventions: Drug: ASP3325
- Japanese male multiple ASP dose-4 (Experimental): ASP3325 will be administered as multiple oral doses with 240 mL of water, three times a day, just after a meal.
  Interventions: Drug: ASP3325
- Japanese male multiple ASP dose-5 (Experimental): ASP3325 will be administered as multiple oral doses with 240 mL of water, three times a day, just after a meal.
  Interventions: Drug: ASP3325
- Japanese female multiple ASP dose-3 (Experimental): ASP3325 will be administered as multiple oral doses with 240 mL of water, three times a day, just after a meal.
  Interventions: Drug: ASP3325
- Japanese female multiple ASP dose-4 (Experimental): ASP3325 will be administered as multiple oral doses with 240 mL of water, three times a day, just after a meal.
  Interventions: Drug: ASP3325
- Japanese female multiple ASP dose-5 (Experimental): ASP3325 will be administered as multiple oral doses with 240 mL of water, three times a day, just after a meal.
  Interventions: Drug: ASP3325
- Japanese male multiple Placebo (Experimental): Placebo will be administered with 240 mL of water, three times a day, just after a meal.
  Interventions: Drug: Placebo
- Japanese female multiple Placebo (Experimental): Placebo will be administered with 240 mL of water, three times a day, just after a meal.
  Interventions: Drug: Placebo
- Japanese male ASP dose-5 before a meal (Experimental): ASP3325 will be administered with 240 mL of water, three times a day, for 2 days.
  Interventions: Drug: ASP3325
- Japanese male ASP dose-5 during a meal (Experimental): ASP3325 will be administered with 240 mL of water, three times a day, for 2 days.
  Interventions: Drug: ASP3325
- Japanese male ASP dose-5 after a meal (Experimental): ASP3325 will be administered with 240 mL of water, three times a day, for 2 days.
  Interventions: Drug: ASP3325

INTERVENTIONS:
Drug: ASP3325
  Arms: Caucasian male single fasted ASP dose-3; Caucasian male single fasted ASP dose-5; Japanese female multiple ASP dose-3; Japanese female multiple ASP dose-4; Japanese female multiple ASP dose-5; Japanese female single fasted ASP dose-3; Japanese female single fasted ASP dose-5; Japanese male ASP dose-5 after a meal; Japanese male ASP dose-5 before a meal; Japanese male ASP dose-5 during a meal; Japanese male multiple ASP dose-3; Japanese male multiple ASP dose-4; Japanese male multiple ASP dose-5; Japanese male single fasted ASP dose-1; Japanese male single fasted ASP dose-2; Japanese male single fasted ASP dose-3; Japanese male single fasted ASP dose-4; Japanese male single fasted ASP dose-5; Japanese male single fasted ASP dose-6; Japanese male single fasted ASP dose-7; Japanese male single fed ASP dose-5
Drug: Placebo
  Arms: Caucasian male single fasted placebo; Japanese female multiple Placebo; Japanese female single fasted placebo; Japanese male multiple Placebo; Japanese male single fasted placebo; Japanese male single fed placebo

SUMMARY:
The objectives of this study are to evaluate the safety and tolerability of a single and multiple oral dose of ASP3325 and to evaluate the effect of administration timing on the pharmacodynamics of ASP3325 orally administered three times a day.

DETAILED DESCRIPTION:
<Part 1: Single ascending dose> Primary objective

* To evaluate the safety and tolerability of a single oral dose of ASP3325 in non-elderly, healthy adult Japanese male and female, and Caucasian male subjects

Secondary objectives

* To evaluate the pharmacokinetics and pharmacodynamics
* To evaluate gender differences in the pharmacokinetics and pharmacodynamics
* To evaluate ethnic differences in the pharmacokinetics and pharmacodynamics between Japanese and Caucasians

<Part 2: Multiple ascending dose> Primary objective

* To evaluate the safety and tolerability of multiple oral doses of ASP3325 in non-elderly, healthy adult Japanese male and female subjects

Secondary objectives

* To evaluate the pharmacokinetics and pharmacodynamics
* To evaluate gender differences in the pharmacokinetics and pharmacodynamics

<Part 3: Evaluation of the effect of administration timing> Primary objective

* To evaluate the effect of administration timing on the pharmacodynamics of ASP3325 orally administered three times a day at different administration timings of 30 minutes before a meal, during a meal, 30 minutes after a meal, and 2 hours after a meal in non-elderly, healthy adult Japanese male subjects in a crossover design

Secondary objective

* To evaluate the safety and pharmacokinetics

ELIGIBILITY:
Inclusion Criteria:

* body weight (at screening)

  * Japanese male: ≥50.0 kg, <80.0 kg
  * Japanese female: ≥40.0 kg, <70.0 kg
  * Caucasian male: ≥50.0 kg, <100.0 kg
* BMI (at screening)

  * Japanese: ≥17.6 kg/m2, <26.4 kg/m2
  * Caucasians: ≥18.5 kg/m2, <30.0 kg/m2
* Ethnicity

  * Japanese: (1) The investigator or subinvestigator will confirm the ethnicity based on appearance (skin color: yellow) and the fact that both parents and four grandparents are of the same race (lineage) based on an interview. (2) The subject has not resided outside Japan for 5 years or longer.
  * Caucasians: (1) The investigator or subinvestigator will confirm ethnicity based on appearance (skin color: white or brown) and the fact that both parents and four grandparents are of the same race (lineage) based on an interview. (2) The subject has not resided outside the subject's own country for 5 years or longer.
* Healthy, as judged by the investigator or subinvestigator based on the results of a medical examination (subjective symptoms and objective findings) and all tests obtained at screening and during the period from hospitalization to immediately before administration.

Exclusion Criteria:

* Received any investigational drugs in other clinical or post-marketing studies within 120 days before the screening or during the period from the screening to hospitalization (Day -2 [Part 1] or Day -3 [Part 2 and Part 3]) or is scheduled to receive any investigational drugs.
* Donated more than or equal to 400 mL of whole blood within 90 days before the screening or during the period from the screening to hospitalization (Day -2 [Part 1] or Day -3 [Part 2 and Part 3]), more than or equal to 200 mL of whole blood within 30 days, or blood components within 14 days before the screening, or is scheduled to donate more than or equal to 400 mL of whole blood or blood components.
* Received medications, vitamins including vitamin D, or supplements including calcium, iron, magnesium, or niacin (nicotinic acid or nicotinamide), or is scheduled to receive medications, within 7 days before hospitalization (Day -2 [Part 1] or Day -3 [Part 2 and Part 3]).
* A deviation from the normal range of blood pressure, pulse rate, body temperature, or standard 12-lead electrocardiogram (ECG) at screening or Day -1.
* Any deviation of the following criteria for laboratory tests at screening or Day -1. The normal ranges specified at the study site or the test/assay organization will be used as the normal ranges in this clinical study.

  * Hematology:

    1. A deviation of +20% from the upper limit or -20% lower limit of the normal range. However, if the WBC is within the normal range, each differential count of leukocytes will be ignored.
  * Biochemistry:

    1. A deviation from the normal range for AST, ALT, Cre, blood glucose, and serum electrolytes (Na, K, Cl, Mg, Ca, and P).
    2. A deviation of +20% from the upper limit or -20% lower limit of the normal range for other parameters than the above. However, the lower limit of the normal range will not be established for parameters for which a deviation from the lower limit is not considered clinically significant (AST, ALT, γ-GTP, T-Bil, D-Bil, I-Bil, ALP, LDH, CK, T-Cho, TG, TBA, BUN, Cre, and UA). TBA and iPTH will only be confirmed by laboratory tests at screening.
  * Urinalysis:

    1. A deviation from the normal range of each test parameter (female subjects in Part 2 who are menstruating at screening may be eligible even if urinary blood is positive).
  * Urinary drug abuse test:

    1. A positive result for benzodiazepines, cocaine-based narcotics, analeptic drugs, cannabis, barbituric acid derivatives, morphine-based narcotics, phencyclidines, or tricyclic antidepressants.
  * Immunological test (at screening only):

    1. A positive result for HBs antigen, HBc antibody, HAV antibody (IgM), HCV antibody, HIV antigen/antibody, or syphilis.
  * Pregnancy test:

    1. Female subjects who tested positive for pregnancy.
* Failure to meet any criteria for 12-lead ECG for QT assessment at screening (Part 1 and Part 2 only).
* Women who are or may be pregnant, lactating mothers, or women who wish to become pregnant during the study period.
* Concurrent or history of drug allergies.
* Upper gastrointestinal disease (e.g. nausea, vomiting, and stomachache) within 7 days before hospitalization (Day -2 [Part 1] or Day -3 [Part 2 and Part 3]).
* Concurrent or previous hepatic disease (e.g. viral hepatitis and drug-induced liver injury).
* Concurrent or previous heart disease (e.g. congestive heart failure, ischemic heart disease, and arrhythmia requiring treatment).
* Concurrent respiratory disease (e.g. bronchial asthma and chronic bronchitis) or previous serious respiratory disease (except for a history of childhood asthma).
* Concurrent gastrointestinal disease (e.g. peptic ulcer and gastroesophageal reflux esophagitis) or previous serious gastrointestinal disease (except for a history of appendicitis).
* Previous operation of gut excision (except for a history of appendectomy).
* Concurrent or previous renal disease (e.g. acute renal failure, glomerulonephritis, and interstitial nephritis; except for a history of calculus).
* Concurrent or previous endocrine disease (e.g. hyperthyroid, hypothyroid, abnormality of growth hormone).
* Concurrent or previous cerebrovascular disorder (e.g. cerebral infarction).
* Concurrent or previous malignant tumor.
* Excessive drinking or smoking habit. [Measure of "excessive"]:

  * Alcohol: ≥45 g/day [a large bottle of beer contains 25 g of alcohol, and 1 gou of Japanese sake contains 22 g of alcohol]
  * Smoking: ≥20 cigarettes/day
* Irregular defecation pattern (less frequent than once a day) (Part 2 and Part 3 only).
* Unable to consume or tolerate phosphorus- and calcium-controlled meals during hospitalization.

Ages: 20 Years to 44 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 124 (Actual)
Dates: Start 2013-07; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Safety developed by adverse events, Part 1 | Up to Day 7 under Fasted and Fed Conditions
Safety developed by adverse events, Part 2 | Up to Day 13
Safety developed by adverse events, Part 3 | Up to Day 8 in Period 4
Safety developed by Vital signs, Part 1 | Up to Day 7
Safety developed by Vital signs, Part 2 | Up to Day 13
Safety developed by Vital signs, Part 3 | Up to Day 8 in Period 4
Safety developed by Laboratory Tests, Part 1 | Up to Day 7 under Fasted and Fed Conditions
Safety developed by Laboratory Tests, Part 2 | Up to Day 13
Safety developed by Laboratory Tests, Part 3 | Up to Day 8 in Period 4
Safety developed by 12-Lead ECG, Part 1 | Up to Day 7 under Fasted and Fed Conditions
  ECG = electrocardiogram
Safety developed by 12-Lead ECG, Part 2 | Up to Day 13
  ECG = electrocardiogram
Safety developed by 12-Lead ECG, Part 3 | Up to Day 8 in Period 4
  ECG = electrocardiogram

SECONDARY OUTCOMES:
12-lead continuous ECG for QT assessment | Up to Day 2 in examination only for administration under fasted condition in Part 1 and Part 2
  ECG: Electrocardiogram
Standard 12-lead ECG for QT assessment | Day -1 ~ 2 in Part 1 and from Day -1 ~1 and Day7~8 in Part 2
  ECG: Electrocardiogram
Plasma concentration of ASP3325 | Day 1, 2, 3 and 4 in Part 1 under Fasted and Fed Conditions, Day 1, 2, 4, 6, 7, 8, 9 and 10 in Part 2, Day 1, 2, 3, 4, 5 in Part 3
Urinary concentration of ASP3325 | Day 1, 2, 3 and 4 in Part 1 under Fasted and Fed Conditions, Day -1, 1, 2, 7, and 8 in Part 2, Day -1, 1, 2, 3, 4, 5 in Part 3
Amount of phosphorus excreted in urine and FEP% | Day 1, 2, 3 and 4 in Part 1 under Fasted Conditions
  FEP% = Fractional Phosphate Excretion
Amount of phosphorus excreted in urine | Day -1, 1, 2, 3, 4, 5, 6, 7, 8, 9, and 10 in Part 2
Amount of calcium excreted in urine | Day -1, 1, 2, 7, 8, 9, and 10 in Part 2
Amount of phosphorus excreted in feces | Day -1, 1, 2, 3, 4, 5, 6, 7, 8, 9, and 10 in Part 2
Amount of calcium excreted in feces | Day -1, 1, 2, 7, 8, 9, and 10 in Part 2
Amount of FEP% | Day -1, 1, 2, 7, 8, 9, and 10 in Part 2
  FEP%：Fractional phosphate excretion
Amount of phosphorus excreted in urine | Day -1, 1, 2, 3, and 4 in Part 3
Amount of calcium excreted in urine | Day -1, 1, 2, 3, and 4 in Part 3
Amount of phosphorus excreted in feces | Day -1, 1, 2, 3, and 4 in Part 3
Amount of calcium excreted in feces | Day -1, 1, 2, 3, and 4 in Part 3
Amount of FEP% | Day -1, 1, 2, 3, and 4 in Part 3
  FEP%: Fractional phosphate excretion

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Astellas Pharma Inc
Locations (1):
- Tokyo, Japan